CLINICAL TRIAL: NCT03475589
Title: A Clinical Study Investigating Adverse Drug Reactions and Their Biomarker Correlations in Stage IV Cancer Patients Following Individualized Therapy of Apatinib
Brief Title: Study on the Adverse Drug Reactions (ADRs) of Apatinib and Their Biomarker Correlations
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Hao Long, Sun Yat-sen University cancer center, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: A2018-002
Record Dates: First submitted 2018-03-18; First posted 2018-03-23 (Actual); Last update posted 2020-05-12 (Actual); Status verified 2020-05

CONDITIONS: Stage IV Cancer
Keywords: apatinib； Adverse drug reactions； gastric cancer; non-small cell lung cancer;breast cancer; ovarian cancer
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms | interventions — apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single group (Other)
  Interventions: Drug: apatinib

INTERVENTIONS:
Drug: apatinib — Patients with advanced (stage IV) gastric cancer, non-small-cell lung cancer (NSCLC), breast cancer or ovarian cancer will be included in this study to receive apatinib treaetment starting from 250 mg Qd and closely monitored for ADRs during apatinib treatment, with dosage adjustment performed as needed to make the treatment tolerable to the patients.

SUMMARY:
The tolerability of apatinib, an effective antiangiogenic agent, varies greatly in patients with stage IV cancer during treatment. This study will include patients with advanced (stage IV) gastric cancer, non-small-cell lung cancer (NSCLC), breast cancer or ovarian cancer, who will be administered apatinib treatment starting from 250 mg Qd and closely monitored for ADRs during the period of apatinib treatment. Meanwhile, relevant assay technologies will be used to precisely detect changes of various biomarkers in the patients treated by apatinib, with the aim of identifying biomarkers related to their prognosis and relevant complications so as to screen out the favored population, establish the drug's indication(s) and reduce relevant side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 and over, male or female;
2. Patients with histologically confirmed advanced (stage IV) gastric cancer, NSCLC, breast cancer or ovarian cancer, who choose monotherapy of oral vascular targeting drug (apatinib) due to intolerability or inappropriateness of other therapies;
3. Presence of measurable lesions (≥10mm on spiral CT scan) subject to RECIST 1.1;
4. Blood pressured controlled at 150/100 mHg following drug administration;
5. An ECOG PS score of between 0 and 1;
6. Findings of hematology and laboratory tests at the baseline that meet the following criteria:

   Hemoglobin ≥80g/L; Absolute neutrophil count (ANC) ≥1.5×10^9/L; Platelets ≥90×10^9/L; ALT/AST ≤ 2.5×ULN; or ALT/AST ≤ 5×ULN for patients with hepatic metastases; Serum total bilirubin ≤1.5×ULN; Serum urea nitrogen and creatinine ≤ 1.5×ULN; Serum albumin ≥30g/L; Coagulation function (INR≤1.5, APTT≤1.5 ULN);
7. A life expectancy of at least 3 months;
8. Subjects who volunteer to participate in this study and have signed the Informed Consent Form (ICF), with good compliance with treatment and follow-up.

Exclusion Criteria:

1. Confirmed allergy to apatinin and or its excipients;
2. Hypertension (high blood pressure) that can not be controlled by drugs;
3. A history of active hemorragge, ulcer, intestinal perforation, intestinal obstruction, or major surgery no older than 30 days;
4. NYHA III-IV heart function, or severe hepatic or renal insufficiency (Grade 4);
5. Presence of multiple factors that affect oral medications, such as difficulty swallowing, nausea, vomiting, chronic diarrhea and intestinal obstruction;
6. Pregnant or lactating women, or women of child-bearing potential who have planned a pregnancy, or male and female patients who do not agree to practice adequate contraception during this study;
7. Patients who have a history of psychotropics abuse and can not quit, or who have mental disorders;
8. Participation in other drug clinical trial within the last 4 weeks;
9. Prior therapy with VEGFR inhibitors such as sorafenib and sunitinib;
10. Presence of comorbidities that seriously affect the patient's safety or ability to complete the study, in the investigator's judgment;
11. Patients who can not tolerate apatinib treatment as judged by the investigator depending on the their medical history;
12. Patients that are considered ineligible for this study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Estimated)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
metastasis | eight weeks
  The patient was diagnosed as recurrence or metastasis according to the computed tomography (CT) scan

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China